CLINICAL TRIAL: NCT03142828
Title: Effect of the Application of Chlorhexidine in the Pillars of Implant Healing to Prevent Plate Accumulation. Controlled Random Blind Clinical Study.
Brief Title: Implant Healing Abutment and Chlorhexidine
Acronym: CHX-HA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Arturo Sánchez-Pérez, Associate professor, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1366/2016
Record Dates: First submitted 2017-03-20; First posted 2017-05-05 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Periimplantitis
Keywords: chlorhexidine, dental implant, in-situ drug delivery,
MeSH Terms: conditions — Peri-Implantitis | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: After the first week, the healling abutment will be randomly distributed in a test group with application of chlorhexidine gel or a control group without the application of the chlorhexidine gel.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blindness performed for patients and for statistical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (clorhexidine gel) (Active Comparator): The healing abutments were covered by a chlorhexidine gel after the first week of the second surgery (2-stage implants).
  Interventions: Drug: Chlorhexidine
- Placebo (Placebo Comparator): The healing abutments were covered without any antiseptic gel after the first week of the second surgery (2-stage implants).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Chlorhexidine — Healing abutment with Clorhexidine
  Other Names: CHX
  Arms: Test (clorhexidine gel)
Other: Placebo — Healing abutment without any antiseptic
  Arms: Placebo

SUMMARY:
The work hyposesis is based on the application of a chlorhexidine gel against the non-application on the healing abutments in patients who have received a submerged titanium implant to check its effect on healing and prevention of bacterial plaque accumulation during a period of 1 month.

DETAILED DESCRIPTION:
Once the implants are integrated, and given the consent, the patients will be operated to connect the healing abutments as they come from the manufacturer (Mozo Grau, Ticare®). Patients will follow the study protocol in 2 arms.

The random distribution is made prior to assignment following the internet program https://www.random.org

ELIGIBILITY:
Inclusion Criteria:

* Good systemic health status (ASA I or II).
* No current pain.
* No use of painkillers or Anti-inflammatory drugs in the prior weeks.
* Older than 18 years.
* Oral hygiene index of ≤ 2 (Löe and Silness).
* A minimum of 2 mm of adhered gum.
* A minimum of 8 mm of vertical bone.
* A minimum of 7 mm of vestibule-lingual bone.
* Scheduled to receive a unitary implant.
* Willing to participate in this controlled study.

Exclusion Criteria:

* Pregnant or nursing women.
* Use of any type of medication that might affect the perception of pain.
* An history of alcohol or drug abuse.
* A requirement for guided regeneration or sinus lifting procedures.
* Failure to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
Degree of inflammation | 1 month after second surgery
  Degree of inflammation was measured using a 4-point Likert scaleInflammation 0 = non-inflamed gingiva with pale pink color. Inflammation 1 = erythematous gingiva without bleeding on manipulation. Inflammation 2 = gingiva with slight bleeding during manipulation during unscrewing or screwing of the abutment. Inflammation 3 = gingiva with heavy bleeding during manipulation during unscrewing or screwing of the abutment.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Sánchez-Pérez, Professor, Principal Investigator — Universidad de Murcia
Locations (1):
- Odontologic Universitary Clinic, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Non-personal data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the publication of the results
Access Criteria: Any interested researcher